CLINICAL TRIAL: NCT01836809
Title: The Impact of Nesiritide on Renal Function After Implantation of the Total Artificial Heart and Left Ventricular Assist Devices
Brief Title: Nesiritide and Renal Function After the Total Artificial Heart
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility for enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM15024
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Congestive Heart Failure; Cardiorenal Syndrome
Keywords: Total Artificial Heart; Left Ventricular Assist Device; Natriuretic peptides; Heart Failure; Cardiorenal Syndrome
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Total Artificial Heart (Experimental): Nesiritide
  Interventions: Drug: nesiritide
- Total Artificial Heart: Placebo (Placebo Comparator): Control arm for subjects receiving the Total Artificial Heart and randomized to receive placebo
  Interventions: Drug: placebo
- LVAD: Nesiritide (Active Comparator): Active arm of the LVAD group
  Interventions: Drug: nesiritide
- LVAD: Placebo (Placebo Comparator): Control arm for subjects receiving LVAD and randomized to placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nesiritide — nesiritide at 0.005 mcg/kg/min without a bolus starting 6 hours after the subject has come off of cardiopulmonary bypass and will continue for 48 hours.
  Other Names: Natrecor
  Arms: LVAD: Nesiritide; Total Artificial Heart
Drug: placebo — placebo bolus starting 6 hours after the subject has come off of cardiopulmonary bypass and will continue for 48 hours.
  Arms: LVAD: Placebo; Total Artificial Heart: Placebo

SUMMARY:
The prevalence of renal dysfunction after implantation of the artificial heart is high. The infusion of exogenous B-type natriuretic peptide (BNP) after implantation of the total artificial heart (TAH) improves renal function in a sustained manner. The renal protective and hormone-modulating effects of nesiritide may be enhanced with ventriculectomy compared to heart failure surgery that leaves the native myocardium intact. The goal of this project is to determine the renal protective effects of nesiritide after implantation of a mechanical device.

DETAILED DESCRIPTION:
This is a randomized, double blinded placebo controlled study that will take place in the Cardiac Surgery Intensive Care Unit, at Virginia Commonwealth University (VCU) Hospital Center.

This study will enroll 20 adult patients who have undergone implantation of a circulatory support device (10 TAH patients, 10 Left ventricular assist device (LVAD) patients). Patients will receive standard postoperative care, including anticoagulation, continuous hemodynamic monitoring with an arterial line and central venous line and hemodynamic support as determine by the cardiac surgery clinical team. We will exclude patients who are receiving renal replacement therapy at the time of device implantation or those that have had previous solid organ transplantation in order to remove the confounding influence of calcineurin inhibitor exposure on renal function. Patient unable to provide informed consent will also be excluded.

Nesiritide Infusion

The patients will be randomized (stratified by device type) to either the study drug (nesiritide at 0.005 mcg/kg/min without a bolus) or placebo. A fixed-dose infusion will be initiated 6 hours after the patients having come off of cardiopulmonary bypass and continued for 48 hours.

Laboratory Measurements

Acute and chronic effects of nesiritide on Glomerular Filtration Rate (GFR) and Renal Plasma Flow (RPF) will be measured by continuous infusion of iothalamate (IOTH) and phenylalanine hydroxylase (PAH), respectively. GFR and RPF will be measured at baseline (-3 to 0 hrs) and at 3 intervals during drug/placebo administration as follows: 0 to 6, 6 to 16 and 16 to 40. Intravenous catheters will be placed as needed for infusion of PAH and IOTH and for timed blood collections.

Urine volume, creatinine, sodium excretion will also be measured. Neurohormones will be measured at all time points 3-6. Plasma renin activity will be measured with an automated chemiluminescent immunoassay (DiaSorin Liaison). Serum aldosterone concentration will be determined by liquid chromatography-mass spectrometry (Agilent, AB Sciex API 5000). Serum BNP concentration will be measured with a sandwich chemiluminescent immunoassay (Siemens Healthcare Diagnostics, ADVIA Centaur BNP immunoassay).

Statistical Analysis Sample size was determined using urine output data from our preliminary observations. Power calculations showed that a total of 10 patients in this two-treatment parallel-design study to have 84 percent power to detect a change in urine output by 75 mL/hr at a two-sided 0.05 significance level (using standard deviation of 35 mL/hr for urine output). Thus 10 patient were included in each device arm of the study.Chi-square analysis was used to compare discrete variables.

A two tailed Student's t-test was used to compare continuous variables. A repeated measures analysis of variance (ANOVA) was used to compare changes in clinical variables laboratory measurements across time points. A P value < 0.05 was considered significant. For individual comparisons post-hoc testing was performed with a paired t-test analysis with Bonferroni correction for 2 comparisons and thus only a P value < 0.025 will considered significant for the repeated measures analyses. A Student 2-tailed paired t test will be used to compare placebo and active drug values for each individual time point.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a total artificial heart (CardioWest) or Left ventricular assist device (HeartMate II)
* Age > 18 years

Exclusion Criteria:

* Previous calcineurin inhibitor (CNI) exposure
* Hemodialysis prior to device implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keyur B. Shah, MD, Principal Investigator — Virginia Commonwealth University Medical Center
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Artificial Heart: Active arm of Total Artificial Heart group
  randomized to receive nesiritide at 0.005 mcg/kg/min without a bolus
- Total Artificial Heart: Placebo: This arm included subject who received a total artificial heart and will be randomized receive placebo
- LVAD: Nesiritide: Active arm of the LVAD group
  randomized to receive nesiritide at 0.005 mcg/kg/min without a bolus
- LVAD: Placebo: This arm will consist of subjects who received an LVAD and will be randomized to placebo
Period: Overall Study
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Started | 0 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total Artificial Heart: Active arm of the Total Artificial Heart group
  randomized to nesiritide
- Total Artificial Heart: Placebo: Total Artificial Heart group
  randomized to placebo
- LVAD: Nesiritide: Active arm of the LVAD group
  randomized to nesiritide
- LVAD: Placebo: Control arm of the LVAD group
  randomized to placebo
- Total: Total of all reporting groups
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
Age, Continuous [Median (Full Range); unit: years] |  |  |  | 59.5 [58 to 61] | 59.5 [58 to 61]
Age, Categorical [Number; unit: participants]
  <=18 years |  |  |  | 0 | 0
  Between 18 and 65 years |  |  |  | 2 | 2
  >=65 years |  |  |  | 0 | 0
Gender [Number; unit: participants]
  Female |  |  |  | 1 | 1
  Male |  |  |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  |  |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Glomerular Filtration Rate
Time Frame: 46 hours
Population: Analysis not done as study was closed early due to futility of reaching enrollment goals in the Total Artificial Heart arm
Groups:
- Total Artificial Heart: Active arm of the Total Artificial Heart group
  randomized to receive nesiritide
- Total Artificial Heart: Placebo: Control arm of the Total Artificial Heart group
  randomized to receive placebo
- LVAD: Nesiritide: Active arm of the LVAD group
  randomized to receive nesiritide
- LVAD: Placebo: Active arm of the LVAD group
  randomized to receive placebo
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Renal Plasma Flow
Time Frame: 46 Hours
Population: as for outcome 1
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Need for Hemodialysis/Renal Replacement Therapy
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Urine Output
Time Frame: 46 Hours
Population: as for outcome 1
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Renal Failure
Time Frame: 46 Hours
Population: as for outcome 1
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Total Diuretic Requirement
Time Frame: 46 Hours
Population: as for outcome 1
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: No unexpected serious adverse events or adverse events were observed
Groups:
- Total Artificial Heart: Active arm of the Total Artificial Heart group
  randomized to receive nesiritide 0.005 mcg/kg/min without bolus
- LVAD: Placebo: Control arm of the LVAD group
  randomized to receive placebo
Arm/Group | Total Artificial Heart | Total Artificial Heart: Placebo | LVAD: Nesiritide | LVAD: Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/2

LIMITATIONS AND CAVEATS:
Enrollment closed. Total Artificial Hearts (TAH) are rarely done as advances with Left Ventricular Assist Devices have improved. We were unable to meet enrollment goal based on the funding timeline due to the lack of TAH's for comparison to LVAD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes